CLINICAL TRIAL: NCT02161185
Title: An Open-Label Safety Study of USL261 in the Outpatient Treatment of Adolescent and Adult Subjects With Seizure Clusters
Brief Title: A Long-term Safety and Tolerability Study of USL261 in Patients With Seizure Clusters
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to slow enrollment. There were no safety concerns.
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P261-408; 2014-001604-22 (EudraCT Number)
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; seizure cluster; acute repetitive seizures; open-label; intranasal Midazolam; USL261; Upsher-Smith
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- USL261 (Other)
  Interventions: Drug: USL261

INTERVENTIONS:
Drug: USL261 — 5 mg, intranasal dose for seizure cluster, may repeat as indicated by protocol
  Other Names: Intranasal Midazolam

SUMMARY:
The purpose of this study is to examine the long-term safety and tolerability of USL261 in the treatment of seizure clusters.

ELIGIBILITY:
Inclusion Criteria:

1. Has a competent, adult caregiver(s) who is able to recognize and observe the subject's seizure cluster episodes
2. Has an established diagnosis of partial or generalized epilepsy that includes all the following:

   * A documented history of seizure clusters lasting a minimum of 10 minutes, seizure cluster pattern is observable, stereotyped, and recognizably different from the subject's other non-cluster seizure activity (if any)
   * A second seizure in the seizure cluster typically occurs within 6 hours from the time of recognition
   * A seizure cluster pattern composed of multiple (≥ 2) partial or generalized seizures
   * A seizure cluster pattern established >3 months before Visit 1
   * A frequency of ≥ 3 stereotyped seizure clusters during the year before Visit 1
   * At least 1 stereotyped seizure cluster occuring ≤ 4 months before Visit 1
3. Currently on a stable regimen of AED(s) that includes a benzodiazepine
4. Weight is 40 kg to 125 kg, inclusive

Exclusion Criteria:

1. Has a neurological disorder that is likely to progress in the next year
2. Has a severe chronic cardio-respiratory disease
3. Has a psychogenic, non-epileptic seizure(s) within the 5 years before Visit 1
4. Has a history of their stereotypical seizure cluster progressing to status epilepticus within 2 years before Visit 1
5. Has a history of acute narrow-angle glaucoma
6. Has had active suicidal plan/intent or active suicidal thoughts in the 6 months before Visit 1 or a suicide attempt in the past 5 years

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TzeChiang Meng, MD, Study Director — Proximagen, LLC
Locations (16):
- United States (16):
  - Tucson, Arizona
  - Fresno, California
  - Ventura, California
  - Aurora, Colorado
  - Port Charlotte, Florida
  - Tampa, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Lexington, Kentucky
  - Saint Paul, Minnesota
  - Reno, Nevada
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Test Dose Phase
Arm/Group | USL261
Started | 7
Completed | 7
Not Completed | 0
Period: Treatment Phase
Arm/Group | USL261
Started (6 of the 7 participants who entered Treatment Phase treated at least one seizure cluster) | 7
Completed (Study discontinued due to poor enrollment) | 0
Not Completed | 7
Not completed — Administrative/Other | 7

BASELINE CHARACTERISTICS:
Arm/Group | USL261
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 27.0 [19 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death, Serious Adverse Events, Treatment Emergent Adverse Events (TEAEs) Leading to Discontinuation
Description: Number of Participants with Death, Serious Adverse Events, Treatment emergent adverse events (TEAEs) leading to subject discontinuation from study
Time Frame: Duration of individual subject participation was open-ended. Study ended early. Longest subject participation approximately 6 months.
Population: Participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | USL261
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Treatment Success
Description: Termination of seizure(s) within 10 minutes and no recurrence within 6 hours after study drug administration. Due to early termination of the study, this data was not analyzed.
Time Frame: as for outcome 1
Population: Not applicable. Only 6 subjects treated at least 1 seizure cluster; of the treated seizure clusters, the majority were in only 2 subjects. Analysis of this endpoint was not performed as the sponsor believed the results would not be interpretable.
Arm/Group | USL261
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Duration of individual subject participation was open-ended. Study ended early. Longest subject participation approximately 6 months.
Description: Treatment emergent
Arm/Group | USL261
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | USL261 (N=7)
Furuncle (Infections and infestations) | 1
Product taste abnormal (General disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Laceration (Injury, poisoning and procedural complications) | 1
Somnolence (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Oxygen saturation decreased (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 1
Lacrimation increased (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination due to poor enrollment leading to small numbers of subjects analyzed for safety. Efficacy was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A manuscript or abstract should not be submitted by investigator(s) for publication or presentation until a New Drug Application is approved by the US FDA or permission is granted in writing by the sponsor.